CLINICAL TRIAL: NCT00777998
Title: Autologous-Allogeneic Tandem Stem Cell Transplantation and Maintenance Therapy With Thalidomide/ DLI for Patients With Multiple Myeloma (MM) and Age < _60 Years: A Phase II-study
Brief Title: Auto-Allo Tandem Stem Cell Transplantation for Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Auto-Allo TSCT in MM
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Stem Cell Transplantation; Thalidomide; DLI
MeSH Terms: conditions — Multiple Myeloma | interventions — Maintenance; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Auto-Allo Tandem Stem cell Transplantation plus maintenance therapy with Thalidomide and DLI
  Interventions: Procedure: Auto-Allo Tandem SCT and maintenance therapy with Thalidomide/ DLI
- B (Active Comparator): Auto-Auto Tandem stem cell Transplantation plus maintenance therapy with Thalidomide
  Interventions: Procedure: auto-auto Tandem stem cell transplantation and maintenance therapy with Thalidomide

INTERVENTIONS:
Procedure: Auto-Allo Tandem SCT and maintenance therapy with Thalidomide/ DLI — *Multiple myeloma
  * -> Induction Therapy (max. 8 cycles)
  * -> Registration of patient, stem cell mobilization, start of donor search
  * -> Melphalan (200mg/qm) plus autologous PBSCT
  * -> 2 months later: Melphalan plus allogeneic PBSCT
  * -> day 120 after allogeneic PBSCT: Thalidomide, 100mg (max. 2 years or until progress or non-tolerable toxicity, respectively)
  * -> day 180 after allogeneic PBSCT (if CsA discontinued): First DLI (1 x 10^6 (MRD) or 5 x 10^5 (MUD) CD3+ cells per kg BW)
  * -> day 250 after allogeneic PBSCT: second DLI (if no signs of GvHD: dose escalation by 0,5 Log)
  * -> Day 320 after allogeneic PBSCT: Third DLI (if no signs of GvHD: dose escalation by 0,5 Log)
  * -> Further DLI depending on MRD-measurement
  Arms: A
Procedure: auto-auto Tandem stem cell transplantation and maintenance therapy with Thalidomide — *Multiple myeloma
  * -> Induction Therapy (max. 8 cycles)
  * -> Registration of patient, stem cell mobilization, start of donor search
  * -> Melphalan (200mg/qm) plus autologous PBSCT
  * -> if no donor available (max 4 weeks after autologous PBSCT) or if patients declines allogeneic PBSCT): 2 months: Melphalan (200mg/qm) plus autologous PBSCT
  * -> day 120 after autologous PBSCT: Thalidomide, 100mg (max. 2 years or until progress or non-tolerable toxicity, respectively)
  Arms: B

SUMMARY:
The present study will be a multicenter, prospective phase II-study investigating safety and efficacy of the combination of auto-allo tandem stem cell transplantation in patients with multiple myeloma and age of >_60 years, followed by maintenance therapy with low-dose Thalidomide and Donor Lymphocyte Infusions.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma Stage II or III acc. to Salmon and Durie
* Patient's age 18-60 years
* Patient's written informed consent
* Women and men capable of reproduction must agree to use adequate contraceptive measures (condom, IUD, oral contraceptives) until three months after termination of treatment
* a maximum of eight chemotherapy cycles prior to registration (CR/ PR/ MR/ or PD)

Exclusion Criteria:

* More than eight chemotherapy cycles prior to registration
* severe irreversible renal, hepatic, pulmonary or cardiac disease, such as

  * total bilirubin, SGPT or SGOT > 3 times upper the normal level
  * Left ventricular ejection fraction < 30 %
  * Creatinine Clearance < 30 ml/min
  * DLCO < 35 % and/or receiving supplementary continuous oxygen
* Positive serology for HIV
* Pregnant or lactating women
* Participation in another trial at the time of registration
* Preceding autologous stem cell transplantation
* age > 61 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2008-10-14 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Event-free survival 4 years after auto-allo/ auto-auto Tandem-SCT. Any of the following will be considered an endpoint event: recurrence or progression of primary disease, disease related mortality, or treatment related mortality. | four years after Tandem stem cell transplantation

SECONDARY OUTCOMES:
Incidence of acute GvHD | day +100 after allogeneic stem cell transplantation
Incidence of chronic GvHD | at one year and at two years after allogeneic stem cell transplantation
Toxicity of conditioning regimen and of maintenance therapy | Throughout conditioning regimen and maintenance therapy
cumulative incidence of relapse | four years after Tandem stem cell transplantation
Disease related mortality | four years after allogeneic stem cell transplantation
Treatment related mortality | four years after allogeneic stem cell transplantation
overall survival | four years after allogeneic stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department for Stem Cell Transplantation
Locations (20):
- Germany (20):
  - Klinikum Augsburg, Augsburg
  - Charité, Berlin
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsklinikum Greifswald, Greifswald
  - Universitätsklinikum Halle (Saale), Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Marburg, Marburg
  - Universitätsklinikum Münster, Münster
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Deutsche Klinik für Diagnostik, Wiesbaden
  - Horst Schmidt Kliniken GmbH, Wiesbaden

REFERENCES:
- [Derived] Kroger N, Wulf G, Hegenbart U, Burchert A, Stelljes M, Gagelmann N, Brecht A, Kaufmann M, Muller L, Ganser A, Wolf D, Bethge W, Bornhauser M, Kiehl M, Wagner EM, Schmid C, Reinhardt HC, Kobbe G, Salwender H, Heinicke T, Kropff M, Heinzelmann M, Ayuk F, Trumper L, Neubauer A, Volp A, Kluychnikov E, Schonland S, Wolschke C. Autologous-allogeneic versus autologous tandem stem cell transplantation and maintenance therapy with thalidomide for multiple myeloma patients under 60 years of age: a prospective, phase II study. Haematologica. 2024 May 1;109(5):1469-1479. doi: 10.3324/haematol.2023.282920. PMID 37941409